CLINICAL TRIAL: NCT01966861
Title: Weaning From Mechanical Ventilation Guided by Lung Ultrasound (Brazilian WEANLUS)
Acronym: WEANLUS-BR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Hospital Sirio-Libanes (Other); University of Sao Paulo (Other); Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Jorge Salluh, MD, PhD, D'Or Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDOR-03-2013
Record Dates: First submitted 2013-10-15; First posted 2013-10-22 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Acute Respiratory Failure
Keywords: mechanical ventilation; weaning; acute respiratory failure; weaning failure; lung ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (No Intervention): Weaning as protcolised by the units' daily practice (SBT)
- Weaning guided by lung ultrasound (Experimental): Predictive early signs of respiratory distress are assessed by lung ultrasound and if found will trigger protocolised intervention (eg- fluid balance,diuretics, thoracocentesis)
  Interventions: Other: weaning guided by LUS (lung ultrasound)

INTERVENTIONS:
Other: weaning guided by LUS (lung ultrasound) — Predictive early signs of respiratory distress are assessed by lung ultrasound (LUS score >14) and if present will trigger protocolised intervention (eg- fluid balance,diuretics, thoracocentesis, antibiotics when required [CPIS>6], hemglobin>8g/dl triggers transfusion)
  Arms: Weaning guided by lung ultrasound

SUMMARY:
The present study aims to evaluate the impact of a weaning strategy based on identification of early signs of respiratory distress by lung ultrasound and the consequent implementation of a "clinical optimization" protocol as compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated >48h

Exclusion Criteria:

* Moderate/Severe COPD
* Spinal cord lesion
* Neuromuscular disease (previous)
* Lung fibrosis
* Tracheostomy
* Heart failure (EF<50%)
* Lung/pleural cancer
* inadequate "window"for LUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Respiratory distress requiring re-intubation or non-invasive ventilation | 48hours

SECONDARY OUTCOMES:
28-day mortality | 28 days
Hospital Mortality | Hospital death/discharge (up to 60 days)
Adverse events | 48h
  Renal dysfunction, complications of thoracocentesis, hydro-electrolite changes, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Jorge IF Salluh, MD, PhD, Principal Investigator — D'Or Institute for Research and Education; Luiz M Malbouisson, MD, PhD, Principal Investigator — University of Sao Paulo; Fabiola Prior, MD, Principal Investigator — University of Sao Paulo; Julio Neves, MD, Principal Investigator — Hospital da Bahia; Jean-Jacques Rouby, MD, Study Chair — Paris University
Locations (1):
- D'OR Institute for Research and Education, Rio de Janeiro, Brazil